CLINICAL TRIAL: NCT01991340
Title: H.E.R.O.S. Study: Observational Study to Assess the Cardiac Safety Profile of Trastuzumab in Patients With HER2-positive Breast Cancer.
Brief Title: H.E.R.O.S. Study: An Observational Study of the Cardiac Safety of Herceptin (Trastuzumab) in Patients With HER2-Positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21975
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the safety of Herceptin (trastuzumab) in patients with HER2-positive breast cancer in routine clinical practice. Eligible patients will be followed for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed HER2-positive breast cancer
* Eligible to receive Herceptin as per Summary of Product Characteristics

Exclusion Criteria:

* Contra-indications according to Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive breast cancer eligible for treatment with Herceptin
Sampling Method: Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to approximately 4.5 years

SECONDARY OUTCOMES:
Incidence of symptomatic congestive heart failure (NYHA class II, III and IV) | up to approximately 4.5 years
Incidence of asymptomatic LVEF decline | up to approximately 4.5 years
Frequency of treatment discontinuations/interruptions | up to approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Algeria (7):
  - Algiers
  - Annaba
  - Blida
  - Mascara
  - Oran
  - Sidi Belabes
  - Tizi Ouzou
- Morocco (5):
  - Agadir
  - Casablanca
  - Fes
  - Marrakesh
  - Rabat